CLINICAL TRIAL: NCT04925401
Title: Evaluation of Knowledge About Fever After Consultation in the Pediatric Emergency Department: Standard Consultation Versus Standard Consultation With Distribution of an Information Leaflet About Fever in Pre-consultation
Brief Title: Evaluation of Knowledge About Fever After Consultation in the Pediatric Emergency Department
Acronym: FEARVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APHP210578; 2021-A00643-38 (Other: ID-RCB Number)
Record Dates: First submitted 2021-05-27; First posted 2021-06-14 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Febrile Illness; Fever; Stress
Keywords: Febrile episode; pediatric; pediatric emergency department; therapeutic education
MeSH Terms: conditions — Fever | interventions — Health

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information brochure Arm (Experimental): The experimental group will receive an information brochure on fever in children and how to deal with a febrile episode and usual medical management.
  Interventions: Behavioral: The Information brochure will be created on the basis of information given by the French pediatric network Courlygone and the French National Authority for Health.
- Habitual care (No Intervention): The control group will receive the usual medical management

INTERVENTIONS:
Behavioral: The Information brochure will be created on the basis of information given by the French pediatric network Courlygone and the French National Authority for Health. — An information brochure on fever in children and how to deal with a paediatric febrile episode and usual medical management.
  Arms: Information brochure Arm

SUMMARY:
The purpose of this study is to evaluate the effect of an information brochure on parent / legal guardians' knowledge of what to do about their child's febrile episode after a pediatric emergency department visit.

Single-center randomized controlled trial.

DETAILED DESCRIPTION:
Fever is a common symptom of viral or bacterial infection in pediatrics. Previous studies using both qualitative and quantitative methods have established that intervention with parents/legal guardians on fever management decreases their worry and anxiety related to their child's occurrence of a febrile episode, limits unwise use of antipyretic medication (Walsh, 2006; Walsh, 2008; Peetom, 2017), but also reduces the use of emergency room or telephone medical consultations (Peetom, 2017).

The majority of visits for febrile conditions in children over 3 months of age are avoidable and do not require emergency and/or hospital care. Mistaken beliefs and lack of knowledge about what to do in the event of a febrile episode lead parents to consult a hospital emergency room for their child, which can have an impact on emergency room overcrowding.

The proportion of emergency room visits for febrile conditions assessed by the Intake and Referral Nurse (IOR) as not requiring urgent care raises questions about parents'/legal guardians' knowledge of fever, its monitoring, and what to do during a febrile episode.

The aim of our study is to evaluate parents' knowledge of fever and the appropriate course of action during a febrile episode in a pediatric emergency department of a Parisian university hospital by comparing standard management practices with the knowledge provided by an information brochure.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age
* Be the parent/legal guardian of a child aged between 3 months and 15 years,
* A child with a fever > 38°celsus on arrival at the emergency room (measured by electronic thermometer rectally for children under 2 years of age or axillary/oral for children over 2 years of age),
* Severity of care rating by the IOA grade 4 (non-emergency care)
* Parent affiliated to a social security system or entitled to it
* Parent under "AME" French social security system
* Parent informed and having signed the consent

Exclusion Criteria

* Parent/legal guardian who does not speak or read French,
* Child with a pathology that does not allow for rectal temperature taking
* Parent/legal guardian with a visual impairment that prevents reading the information note and/or the information brochure.
* Parent / legal guardian under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with correct answer to question about management of a paediatric febrile episode. | 1 day
  Number of correct answers to question n°7 (what to do during a febrile episode) of the questionnaire

SECONDARY OUTCOMES:
Number of participants with correct answer to question n°1 about knowledge about paediatric febrile episode | 1 day
  Answer to question n°1, 2, 3, 4, 5, 6, 8, 9 & 10. Number of participants with correct answers, between the two arms
Number of participants with correct answer to question n°2 about knowledge's about paediatric febrile episode | 1 day
  Answer to question n° 2. Number of participants with correct answers, between the two arms. Factors associated with a high number of correct responses: age of child, age of legal guardian, socio-professional category, child's place in sibling group, child's medical follow-up.
Number of participants with correct answer to question n°3 about knowledge's about paediatric febrile episode | 1 day
  Answer to question n° 3. Number of participants with correct answers, between the two arms.
Number of participants with correct answer to question n°4 about knowledge's about paediatric febrile episode | 1 day
  Answer to question n° 4. Number of participants with correct answers, between the two arms.
Number of participants with correct answer to question n°5 about knowledge's about paediatric febrile episode | 1 day
  Answer to question n° 5. Number of participants with correct answers, between the two arms.
Number of participants with correct answer to question n°6 about knowledge's about paediatric febrile episode | 1 day
  Answer to question n° 6. Number of participants with correct answers, between the two arms.
Number of participants with correct answer to question n°8 about knowledge's about paediatric febrile episode | 1 day
  Answer to question n° 8. Number of participants with correct answers, between the two arms.
Number of participants with correct answer to question n°9 about knowledge's about paediatric febrile episode | 1 day
  Answer to question n° 9. Number of participants with correct answers, between the two arms.
Number of participants with correct answer to question n°10 about knowledge's about paediatric febrile episode | 1 day
  Answer to question n° 10. Number of participants with correct answers, between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Hélène CHAPPUY, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- APHP Assistance Publique des Hôpitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmitt BD. Fever phobia: misconceptions of parents about fevers. Am J Dis Child. 1980 Feb;134(2):176-81. PMID 7352443
- [Background] Poirier MP, Davis PH, Gonzalez-del Rey JA, Monroe KW. Pediatric emergency department nurses' perspectives on fever in children. Pediatr Emerg Care. 2000 Feb;16(1):9-12. doi: 10.1097/00006565-200002000-00003. PMID 10698135
- [Background] Burokiene S, Kairiene I, Stricka M, Labanauskas L, Cerkauskiene R, Raistenskis J, Burokaite E, Usonis V. Unscheduled return visits to a pediatric emergency department. Medicina (Kaunas). 2017;53(1):66-71. doi: 10.1016/j.medici.2017.01.003. Epub 2017 Jan 31. PMID 28233682
- [Background] Bereznicki BJ, Tucker MG, Beggs SA, Zosky GR, Bereznicki LR. Emergency department presentations of febrile children to an Australian public hospital. J Paediatr Child Health. 2018 Dec;54(12):1308-1313. doi: 10.1111/jpc.14071. Epub 2018 Jun 6. PMID 29874409
- [Background] Enarson MC, Ali S, Vandermeer B, Wright RB, Klassen TP, Spiers JA. Beliefs and expectations of Canadian parents who bring febrile children for medical care. Pediatrics. 2012 Oct;130(4):e905-12. doi: 10.1542/peds.2011-2140. Epub 2012 Sep 10. PMID 22966028
- [Background] Betz MG, Grunfeld AF. 'Fever phobia' in the emergency department: a survey of children's caregivers. Eur J Emerg Med. 2006 Jun;13(3):129-33. doi: 10.1097/01.mej.0000194401.15335.c7. PMID 16679875
- [Background] Morrison AK, Chanmugathas R, Schapira MM, Gorelick MH, Hoffmann RG, Brousseau DC. Caregiver low health literacy and nonurgent use of the pediatric emergency department for febrile illness. Acad Pediatr. 2014 Sep-Oct;14(5):505-9. doi: 10.1016/j.acap.2014.05.001. Epub 2014 Jun 16. PMID 24942934
- [Background] Walsh A, Edwards H. Management of childhood fever by parents: literature review. J Adv Nurs. 2006 Apr;54(2):217-27. doi: 10.1111/j.1365-2648.2006.03802.x. PMID 16553708
- [Background] Walsh A, Edwards H, Fraser J. Parents' childhood fever management: community survey and instrument development. J Adv Nurs. 2008 Aug;63(4):376-88. doi: 10.1111/j.1365-2648.2008.04721.x. PMID 18727765
- [Background] Peetoom KK, Smits JJ, Ploum LJ, Verbakel JY, Dinant GJ, Cals JW. Does well-child care education improve consultations and medication management for childhood fever and common infections? A systematic review. Arch Dis Child. 2017 Mar;102(3):261-267. doi: 10.1136/archdischild-2016-311042. Epub 2016 Jul 18. PMID 27432451
- [Background] Considine J, Brennan D. Effect of an evidence-based education programme on ED discharge advice for febrile children. J Clin Nurs. 2007 Sep;16(9):1687-94. doi: 10.1111/j.1365-2702.2006.01716.x. PMID 17727587
- [Background] Monsma J, Richerson J, Sloand E. Empowering parents for evidence-based fever management: An integrative review. J Am Assoc Nurse Pract. 2015 Apr;27(4):222-9. doi: 10.1002/2327-6924.12152. Epub 2014 Jul 25. PMID 25066313
- [Background] Broome ME, Dokken DL, Broome CD, Woodring B, Stegelman MF. A study of parent/grandparent education for managing a febrile illness using the CALM approach. J Pediatr Health Care. 2003 Jul-Aug;17(4):176-83. doi: 10.1067/mph.2003.4. PMID 12847427
- [Background] Baker MD, Monroe KW, King WD, Sorrentino A, Glaeser PW. Effectiveness of fever education in a pediatric emergency department. Pediatr Emerg Care. 2009 Sep;25(9):565-8. doi: 10.1097/PEC.0b013e3181b4f64e. PMID 19755888